CLINICAL TRIAL: NCT02764801
Title: 2D and 4D Contrast-enhanced Ultrasound Evaluation of Hepatocellular Carcinoma Chemoembolization
Brief Title: Contrast-enhanced Ultrasound Evaluation of Chemoembolization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: University of California, San Diego (Other); Vanderbilt University Medical Center (Other); National Institutes of Health (NIH) (NIH); Lantheus Medical Imaging (Industry); GE Healthcare (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15F.579; R01CA194307 (NIH); JT 8348 (Other: JeffTrial Number)
Record Dates: First submitted 2016-04-21; First posted 2016-05-06 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma; Chemoembolization, Therapeutic
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Contrast ultrasound arm (Experimental): Patients receiving contrast-enhanced ultrasound for diagnosis of chemoembolization response.
  Interventions: Drug: Ultrasound contrast agent (Contrast-enhanced ultrasound); Device: Logiq E9 Scanner (Contrast-enhanced ultrasound)

INTERVENTIONS:
Drug: Ultrasound contrast agent (Contrast-enhanced ultrasound) — Intravenous injection of ultrasound contrast agent followed by saline flush though an angiocatheter in the arm or hand.
  Other Names: Definity (Lantheus Medical Imaging); Microbubble contrast agent
Device: Logiq E9 Scanner (Contrast-enhanced ultrasound) — Ultrasound scanning using a commercial scanner with a C1-5-D broad-spectrum convex transducer followed by a RAB2-5-D broad-spectrum real-time 4D transducer.
  Other Names: Ultrasound Scanner

SUMMARY:
The primary objective of this trial is to evaluate the sensitivity and specificity of 2D and 4D contrast enhanced ultrasound for monitoring transarterial chemoembolization (TACE) response 1-2 weeks and 1 month post treatment as an alternative to contrast-enhanced magnetic resonance (MRI) or computed tomography (CT) imaging

DETAILED DESCRIPTION:
This is an open-label, non-randomized trial that will be conducted at three clinical sites. The subject population will be patients undergoing transarterial chemoembolization for the treatment of hepatocellular carcinoma (HCC) at Thomas Jefferson University, The University of California, San Diego, and Vanderbilt University. Patients will receive a contrast-enhanced ultrasound (CEUS) exam the morning prior to embolization, approximately one week post-embolization, and at their one month MRI follow up (scheduled as part of their clinical standard of care).

This trial will consist of up to 210 adults (70 per institution) undergoing transarterial chemoembolization for the treatment of HCC split evenly between Thomas Jefferson University, The University of California, San Diego, and Vanderbilt University.

Patients will be identified and consecutively approached from each institution's Hepatology / Transplant Surgery and Interventional Radiology practices (by each site's Hepatology or Interventional Radiology co-investigators). An investigator or research coordinator will explain the study to the patient. The patient will be given time to consider the risks and benefits of the study and to ask questions about participation. A consent form will be reviewed with the patient. A full history and physical examination will be obtained from the patient's referring physician. If the subject is a woman of childbearing potential, she will have a urine pregnancy test prior to each CEUS study (the results of which will be made available to the subject prior to study initiation). In the event a patient presents with a lesion that is expected to be difficult to view on ultrasound (for example, smaller lesions located high on the liver dome), grayscale ultrasound imaging will quickly be performed to ensure the lesion is visible on ultrasound and that the patient is suitable for study inclusion.

Patients will undergo a total of three separate CEUS exams. These exams will consist of the baseline study the morning prior to TACE therapy, a study 1-2 weeks post treatment that will coincide with clinical post-procedure follow-up by the interventional radiologist, and a study approximately one month post treatment when patients return for clinically scheduled CE-CT/MRI follow-up. If the patient fails to show up for the 1-2 week CEUS exam, they will not be excluded from the final ultrasound exam. Procedures and equipment for this trial will be used in accordance with standard clinical protocols and good clinical practices already in place at our hospitals.

The first three cases at each institution (baseline and at least one follow-up) will be performed under the guidance of at least one of the study PIs to ensure standardization amongst all three sites. The ultrasound examinations will be performed by a qualified sonographer. Efforts will be made to have all CEUS scans performed by the same dedicated sonographer, enabling us to evaluate operator dependence. During the ultrasound examination, the patient will be asked to lie in the supine position and a 20-22 gauge cannula will be placed in a superficial vein (preferably an antecubital vein). Ultrasound imaging will be performed using a state of the art Logiq E9 scanner with C1-5-D broad-spectrum convex transducer and a RAB2-5-D broad-spectrum real-time 4D transducer (GE Healthcare, Wauwatosa, WI). As part of this study, the investigators have budgeted for the purchase of 3 4D probes (not routinely available in clinical practice) and the installation of GE's ultrasound volumetric and contrast imaging packages that provide 2D and 4D CEUS capabilities. In the event the patient has multiple lesions scheduled for treatment, up to 2 lesions will be imaged independently on CEUS. Patients will first undergo 2D baseline imaging. B-mode measurements and sweeps of the lesion in the transverse and sagittal planes will be performed, followed by standard power Doppler imaging (PDI). Following baseline imaging, patients will receive a bolus IV injection of up to 0.6 ml of Definity, followed by a 10 cc saline flush. Since Definity is currently only approved for echocardiography, the investigators have applied to the FDA for an investigational new drug application for CEUS evaluation of TACE.

All CEUS imaging will be performed using the dual B-mode (used to locate anatomical features) and nonlinear contrast (to identify the ultrasound contrast agent) imaging mode. A low mechanical index (< 0.1) will be used to minimize microbubble destruction during imaging. The standard nonlinear imaging frequency pairings in the contrast imaging software will be used (transmitting at 2 MHz, receiving at the 4 MHz harmonic), and gain settings will be adjusted to minimize nonlinear signals prior to contrast injection. Additionally, the focal zone will be placed at the approximate depth of the lesion to maximize the generation of nonlinear signals during CEUS. During the first contrast injection, 2D CEUS will be performed using the coded harmonics nonlinear imaging package on the unit. The approximate tumor mid-line will be imaged until homogenous liver enhancement is achieved (approximately 45 seconds post injection), followed by imaging sweeps through the tumor. Sweeps will then be acquired in the sagittal plane, before returning to the original plane. Imaging will be continued until contrast washout is observed (approximately 3-4 minutes), after which data will be digitally stored for later review. A fifteen minute wait period will be observed between injections to allow for complete ultrasound contrast agent clearance. A region of interest encompassing the entire tumor volume and margin will then be selected in 4D mode. Baseline imaging of the tumor will be repeated in 4D mode in grayscale B-mode. A second bolus injection of up to 0.6 ml Definity followed by 10 cc saline flush will again be administered during continuous tumor imaging in 4D, which uses the machine's coded harmonics package. Data will be obtained until contrast washout is observed and then digitally stored in digital imaging and communications in medicine (DICOM) format for later review.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 21 years of age
* Patient capable of making informed decisions regarding his/her treatment
* Scheduled for TACE treatment of a HCC mass (lesions reported as Liver Imaging Reporting and Data Systems 4B or 5 or Organ Procurement and Transplantation Network 5a or 5b)
* Negative pregnancy test in a female of child-bearing age.
* Have an HCC mass viewable on grayscale B-mode ultrasound.

Exclusion Criteria:

* Females who are pregnant or nursing.
* Patients not eligible or scheduled for TACE of a HCC mass.
* Patients who have received an investigational drug in the 30 days before study drug administration, or will receive one within 72 h after their final CEUS exam.
* Patients who have received prior radioembolization (Y90) of the lesion of interest.
* Patients with known or suspected cardiac shunts.
* Patients with pulmonary hypertension or unstable cardiopulmonary conditions.
* Patients who are medically unstable, patients who are seriously or terminally ill, and patients whose clinical course is unpredictable. For example:
* Patients with unstable occlusive disease (e.g., crescendo angina)
* Patients with clinically unstable cardiac arrhythmias
* Patients with uncontrolled congestive heart failure (NYHA Class IV)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2016-04; Primary Completion 2021-12 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Eisenbrey, PhD, Principal Investigator — Thomas Jefferson University
Locations (3):
- United States (3):
  - University of California, San Diego, La Jolla, California
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaw CM, Eisenbrey JR, Lyshchik A, O'Kane PL, Merton DA, Machado P, Pino L, Brown DB, Forsberg F. Contrast-enhanced ultrasound evaluation of residual blood flow to hepatocellular carcinoma after treatment with transarterial chemoembolization using drug-eluting beads: a prospective study. J Ultrasound Med. 2015 May;34(5):859-67. doi: 10.7863/ultra.34.5.859. PMID 25911704
- [Background] Kono Y, Lucidarme O, Choi SH, Rose SC, Hassanein TI, Alpert E, Mattrey RF. Contrast-enhanced ultrasound as a predictor of treatment efficacy within 2 weeks after transarterial chemoembolization of hepatocellular carcinoma. J Vasc Interv Radiol. 2007 Jan;18(1 Pt 1):57-65. doi: 10.1016/j.jvir.2006.10.016. PMID 17296705
- [Derived] Savsani E, Shaw CM, Forsberg F, Wessner CE, Lyshchik A, O'Kane P, Liu JB, Balasubramanya R, Roth CG, Naringrekar H, Keith SW, Tan A, Anton K, Bradigan K, Civan J, Schultz S, Shamimi-Noori S, Hunt S, Soulen MC, Mattrey RF, Kono Y, Eisenbrey JR. Contrast-enhanced US Evaluation of Hepatocellular Carcinoma Response to Chemoembolization: A Prospective Multicenter Trial. Radiology. 2023 Oct;309(1):e230727. doi: 10.1148/radiol.230727. PMID 37847138
- See also: Pubmed Abstract — https://www.ncbi.nlm.nih.gov/pubmed/25911704
- See also: Pubmed Abstract — https://www.ncbi.nlm.nih.gov/pubmed/17296705

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Contrast Ultrasound Arm
Started | 131
Completed | 103
Not Completed | 28

BASELINE CHARACTERISTICS:
Arm/Group | Contrast Ultrasound Arm
Number analyzed (Participants) | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 131
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 110
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 78
  More than one race | 0
  Unknown or Not Reported | 21
Region of Enrollment [Number; unit: participants]
  United States | 131

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Correctly Identified as Requiring Tumor Re-treatment Two Weeks After Initial Chemoembolization
Description: The ability of contrast-enhanced ultrasound to detect residual disease (and thereby need for tumor re-treatment) will be determined 1-2 weeks post chemoembolization.
Time Frame: Percentage of patients correctly identified as requiring re-treatment will be identified 1-2 weeks after the subject's chemoembolization procedure
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Contrast Ultrasound Arm
Number analyzed (Participants) | 103
percentage | 94 [88 to 97]

2. Primary Outcome: Percentage of Patients Correctly Identified as Requiring Tumor Re-treatment One Month After Initial Chemoembolization
Description: The ability of contrast-enhanced ultrasound to detect residual disease (and thereby need for tumor re-treatment) will be determined 1 month post chemoembolization.
Time Frame: Percentage of patients correctly identified as requiring re-treatment will be identified 1 month after the subject's chemoembolization procedure
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Contrast Ultrasound Arm
Number analyzed (Participants) | 103
percentage | 91 [84 to 95]

ADVERSE EVENTS:
Time Frame: 5 years
Description: Unlikely patients will die from imaging study
Arm/Group | Contrast Ultrasound Arm
All-Cause Mortality (participants affected / at risk) | 35/103
Serious Adverse Events (participants affected / at risk) | 4/103
Other Adverse Events (participants affected / at risk) | 4/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contrast Ultrasound Arm (N=103)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
episodic atrial fibrillation (Cardiac disorders) | 1 (1)
esophageal variceal bleeding (Respiratory, thoracic and mediastinal disorders) | 1 (1)
late dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contrast Ultrasound Arm (N=103)
nausea/vomiting (Gastrointestinal disorders) | 1 (103)
IV infiltration (Product Issues) | 1 (103)
post-embolization syndrome (General disorders) | 2 (103) — fever, chills, weakness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT02764801/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT02764801/ICF_001.pdf